CLINICAL TRIAL: NCT00498667
Title: Evaluation of the Prognostic Value of Early Interim PET/CT for Prediction of Progression Free Survival of Patients With Aggressive B Cells Non Hodgkin Lymphoma
Brief Title: The Prognostic Value of Interim PET/CT After 2 Cycles of Chemotherapy in Predicting Progression of Non Hodgkins Lymphoma
Status: Withdrawn | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, e_dann, Prof Eldad Dann, Rambam Health Care Campus
Other Study IDs: cc-NHL2615_CTIL
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Lymphoma; Large Cell (Diffuse) With Small Cell, Diffuse
Keywords: PET/CT; Aggressive non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — no biopsies are to be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT: all patients with aggressive lymphoma who had a baseline and interim pet/ct study

SUMMARY:
A retrospective analysis will be performed regarding the usefulness of PET/CT performed following 2 cycle of chemotherapy in evaluation of progression, free survival and overall survival of patients with aggressive non Hodgkin Lymphoma.

DETAILED DESCRIPTION:
Patients who were treated for aggressive non-Hodgkin lymphoma with adriamycin containing regimen, CHOP and High dose CHOP with or without rituximab were evaluated post 2 cycles of chemotherapy to rule out disease progression . Currently a retrospective evaluation of PET/CT as a predictive value for progression free survival and overall survival is evaluated

ELIGIBILITY:
Inclusion Criteria:

* aggressive non-Hodgkin lymphoma b cells
* age 18-70
* bilirubin less then 2
* creatinine less then 2
* Pet/CT performed post 2 cycles

Exclusion Criteria:

* no PET/CT post 2 cycles performed
* bilirubin >2
* creatinine more then 2
* HIV positivity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with agressive non hodgkin lymphoma who had interim pet/ct during therapy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
progression free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eldad J Dann, MD, Principal Investigator — RAMBAM health care campus,Rappaport faculty of medicine Technion Israel Technical institute
Locations (1):
- RAMBAM health care Campus, Haifa, Israel